CLINICAL TRIAL: NCT03734861
Title: A Prospective, Randomized, Controlled Study to Assess Medication Adherence in Children With Asthma Managed on BreatheSmart and Feedback
Brief Title: The Study is Enrolling Kids From 8 to 17 Years Old. The BreathSmart Device Attaches to the Inhaler to Measure Adherence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-043
Record Dates: First submitted 2018-08-30; First posted 2018-11-08 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two arms:
  1. BreathSmart system
  2. Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BreatheSmart System (Experimental): * BreatheSmart mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor real-time adherence and to provide targeted outreach to children with low adherence (intervention arm)
  Interventions: Device: BreatheSmart System
- Standard of Care (Active Comparator): These patients are reminded to adhere to the prescribed standard of care therapy provided by their clinician during their clinical encounters and when the family calls to report an illness.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: BreatheSmart System — * BreatheSmart System: a mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor adherence
  Arms: BreatheSmart System
Other: Standard of Care — These patients are reminded to adhere to the prescribed standard of care therapy provided by their clinician during their clinical encounters and when the family calls to report an illness.
  Arms: Standard of Care

SUMMARY:
Non-adherence to controller medication is a common problem in children with Asthma, resulting in overuse of reliever medication, increased asthma symptoms, more frequent Asthma attacks, and increased emergency room visits and hospital admissions. Additionally, current absence of a gold standard to measure adherence forces clinicians and researchers to rely on patient-self report, which is notoriously inaccurate, to support clinical decision making. Many young patients suffer from both intentional and non-intentional non-adherence, thus an appropriate intervention must address both types. Current studies using electronic monitoring devices (EMDs) primarily focus on non-intentional non-adherence through reminder systems and thus are limited in their ability to engage patients for long-term behavior change.

This trial addresses an important knowledge gap by evaluating whether EMDs with a combination of reminder system and patient education can prove to be effective in increasing adherence rates and can be used in clinical practice to achieve better asthma control and outcomes through improved patient and clinician engagement.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study of children with persistent asthma who are managed on daily inhaled corticosteroids (ICS). 75 children will be randomized 2:1 into one of two arms:

* 50 children will be randomized to BreatheSmart, comprised of:

  * BreatheSmart mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor real-time adherence and to provide targeted outreach to children with low adherence (intervention arm)
* 25 children will be randomized to "standard of care"(control arm). These patients are reminded to adhere to the prescribed standard of care therapy provided by their clinician during their clinical encounters and when the family calls to report an illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 17
* Diagnosis of persistent asthma
* Prescribed an inhaled corticosteroid (ICS) for at least one month prior to enrollment
* Use of a pressurized metered dose inhaler (pMDI) compatible with the Cohero mHealth Herotracker (See Appendix)
* Parent/child possess a compatible smartphone (iOS 8.0 or higher)
* English or Spanish speaking

Exclusion Criteria:

* Presence of another chronic lung disease or condition such as cystic fibrosis, interstitial lung disease, chronic lung disease of prematurity, recurrent aspiration, or presence of tracheostomy
* Presence of other chronic medical condition such as congenital heart disease or immunodeficiency
* Presence of other comorbidities that, in the opinion of the investigator, will interfere with collection of study procedures, or limits life expectancy to < 1 year
* Currently pregnant or planning to become pregnant during the trial period

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tregony Simoneau, MD, Principal Investigator — Connecticut Childrens Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
NA we are not planning on sharing the data

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- [Derived] Hollenbach J, Simoneau T, Sun Y, Becene I, Almeida S, Langton C, Flores G. Design, methods, and baseline characteristics of a pilot, randomized, controlled trial of the effects of an electronic monitoring device on medication adherence in children with asthma. Contemp Clin Trials Commun. 2021 Feb 6;21:100706. doi: 10.1016/j.conctc.2021.100706. eCollection 2021 Mar. PMID 33644492

RESULTS

PARTICIPANT FLOW:
Groups:
- BreatheSmart System: * BreatheSmart mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor real-time adherence and to provide targeted outreach to children with low adherence (intervention arm)
  * BreatheSmart System: a mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor adherence
Period: Overall Study
Arm/Group | BreatheSmart System | Standard of Care
Started | 50 | 25
Completed | 50 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BreatheSmart System: * BreatheSmart mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor real-time adherence and to provide targeted outreach to children with low adherence (intervention arm)
  BreatheSmart System: ○ BreatheSmart System: a mobile application that tracks medication usage and sends real time reminders
  * HeroTracker sensor that counts dosage and monitors real-time medication adherence
  * CoheroConnect provider portal that allows the Investigator to monitor adherence
- Total: Total of all reporting groups
Arm/Group | BreatheSmart System | Standard of Care | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (3) | 11.7 (2.8) | 12 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 40
  Male | 24 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 13 | 34
  Not Hispanic or Latino | 29 | 12 | 41
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 25 | 75
Proportion of days covered (PDC) [Mean (Standard Deviation); unit: proportion of days] — The primary outcome is medication adherence as measured using pharmacy refills. Medication adherence as measured by pharmacy refills was calculated using proportion of days covered (PDC), a validated method of calculating adherence, defined as a ratio of the sum of unique days supplied based on refills over the total number of days in the assessed period. For baseline adherence, PDC was assessed over a six-month period prior to the enrollment date.
  proportion of days | 0.41 (0.30) | 0.41 (0.27) | 0.41 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered (PDC)
Description: Medication adherence among children using BreatheSmart with feedback (intervention) compared to control group (standard of care) at 6 months. The primary outcome was medication adherence as measured using pharmacy refill. Medication adherence as measured by pharmacy refills was calculated using proportion of days covered (PDC), a validated method of calculating adherence, defined as a ratio of the sum of unique days supplied based on refills over the total number of days in the assessed period.
Time Frame: 6 months post start of intervention
Population: Participants in the BreatheSmart arm (intervention) received the EMD, app, and reminder notifications. Participants in the control group continued to receive routine clinical care. They were reminded to adhere to prescribed therapy during their clinical encounters
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 25
proportion of days | 0.39 (0.34) | 0.33 (0.30)

2. Secondary Outcome: Asthma Control Test
Description: The Asthma control Test (ACT) assess a patient's level of asthma control based on responses to 5 symptom-related questions over the past 4 weeks. Respondents must select a number on a 5-point likert scale (1-5) for each item. The response to each question is summed, ranging from 5-25. Scores of 19 or less indicate poorly controlled asthma. Higher scores mean better asthma control.
Time Frame: 6 months post start of intervention
Population: Participants in the intervention group received an electronic monitoring device (Herotracker), which is synced to the BreathSmart mobile app, designed to send reminder notifications to participants, and are able to collect medication adherence data. Participants are able to track and review their medication adherence using the app. Participants in the control group continued to receive routine clinical care. They were reminded to adhere to prescribed therapy during their clinical encounters.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 25
score on a scale
  ACT baseline | 18.9 (4.5) | 17.9 (5.5)
  ACT 3 months | 21.2 (3.7) | 20 (3.4)
  ACT 6 months | 19.7 (3.1) | 17.9 (5.6)

3. Secondary Outcome: FEV1% Predicted
Description: The percent predicted forced expiratory volume in 1 second (FEV1) were evaluated at baseline, 3-months, and 6-months.
Time Frame: Baseline to 6 months
Population: Participants in both arms performed spirometry during clinic visits
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 23
percentage of predicted FEV1
  Baseline | 89.7 (18.2) | 92.4 (15)
  3-months | 86.5 (12.9) | 99.7 (17.8)
  6-months | 90.5 (16.3) | 103.6 (14.8)

4. Secondary Outcome: Changes in Medication Adherence and Lung Function
Description: The correlation between changes in medication adherence and changes in FEV1 percent predicted.
  FEV1 is forced expiratory volume in 1 second is the maximum amount of air that a subject can forcibly expel during the first second following maximal inhalation. FEV1 can be useful to categorize the severity of asthma. Expressing FEV1 as a percentage of the predicted value in a patient is means by which to express this severity.
Time Frame: Baseline to 6 months post start of intervention
Population: The analysis population was comprised of children enrolled in either the control (standard of care) arm or the intervention (Breathesmart, HeroTracker) arm.
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 25
Spearman's correlation coefficient
  FEV1% predicted | 0.221 | 0.283
  FEV1/FVC | -0.081 | 0.174

5. Secondary Outcome: Number of Participants With Visits to ER for Asthma
Description: The overall number of participant-reported provider visits for asthma healthcare utilization (e.g. number of self-reported exacerbations leading to ER visits)
Time Frame: Baseline to 6 months post start of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 25
Participants
  ED visits 3 months | 0 | 1
  ED visits 6 months | 3 | 3

6. Secondary Outcome: Number of Missed Days of School
Description: Average number of days missed from school in the past 30 days
Time Frame: Last 30 days from baseline visit and last 30 days from 6-month follow-up visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | BreatheSmart System | Standard of Care
Number analyzed (Participants) | 50 | 25
days
  Past 30 days from Baseline | 1.12 (1.9) | 1.04 (1.8)
  Past 30 days from 6-month follow-up | 2.1 (1.5) | 3.3 (3.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | BreatheSmart System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 3/50 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BreatheSmart System (N=50) | Standard of Care (N=25)
Caregiver-reported emergency department visit for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
The intervention sample size was limited by the number of EMDs provided by CoHero. In addition, EMD adherence rates cannot directly be compared between the intervention and control groups because of the study design. Furthermore, at the initiation of the study, CoHero had not designed the BreatheSmart app for compatibility with Android smartphones. Thus, a significant proportion of potentially eligible children were18 excluded because of Android phone ownership.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03734861/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03734861/ICF_002.pdf